CLINICAL TRIAL: NCT03144453
Title: Recovery From Anesthesia After Robotic Assisted Radical Cystectomy. Two Different Reversal of Neuromuscular Blockade
Brief Title: Recovery From Anesthesia After Robotic Assisted Radical Cystectomy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Regina Elena Cancer Institute (Other)
Responsible Party: Principal Investigator, Ester Forastiere, MD, Regina Elena Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CE/2288
Record Dates: First submitted 2017-05-03; First posted 2017-05-08 (Actual); Last update posted 2019-01-28 (Actual); Status verified 2019-01

CONDITIONS: Anesthesiology Management
Keywords: Curare; Robotic surgery
MeSH Terms: interventions — Neostigmine; Atropine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Sugammadex (Experimental): The patients received sugammadex as neuromuscular blockade reversal
  Interventions: Drug: Sugammadex Injectable Product
- Standard (Active Comparator): The patients received neostigmine + atropine as neuromuscular blockade reversal
  Interventions: Drug: Neostigmine, Atropine

INTERVENTIONS:
Drug: Sugammadex Injectable Product — Patients receive sugammadex at the end of the surgery
  Arms: Sugammadex
Drug: Neostigmine, Atropine — Patients receive neostigmine+atropine at the end of the surgery
  Arms: Standard

SUMMARY:
Robot-assisted radical cystectomy (RARC) requires specific surgical conditions: steep Trendelenburg position, prolonged pneumoperitoneum, effective neuromuscular block until the final stages of surgery. The aim of this study was to evaluate the quality of awakening in two groups of patients undergoing different combinations of curarization/reversal.

ELIGIBILITY:
Inclusion Criteria:

* ASA (american society of anesthesiologists) score ≤ III
* Patients underwent robotic assisted cystectomy

Exclusion Criteria:

* Cerebrovascular disease
* BMI (body mass index) ≥ 30

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-05-02 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Time to discharge from recovery room | Up to 240 Minutes After recovery
  Time between reversal administration and discharge from the recovery room

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Ester Forastiere, Rome, RM
  - Regina Elena Cancer Institute, Rome, RM